CLINICAL TRIAL: NCT02092259
Title: A Multi-Site Clinical Evaluation of the ARIES Norovirus Assay in Patients With Signs and Symptoms of Acute Gastroenteritis
Brief Title: A Multi-Site Clinical Evaluation of the ARIES Norovirus Assay
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Luminex Corporation (Industry)
Responsible Party: Sponsor
Organization: Luminex Molecular Diagnostics (Industry)
Other Study IDs: LMA-NOR-01-CS-001
Record Dates: First submitted 2014-03-17; First posted 2014-03-20 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-06

CONDITIONS: Acute Gastroenteritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool
Oversight: Data Monitoring Committee: No

SUMMARY:
The ARIES Norovirus Assay is a real-time PCR based qualitative in vitro diagnostic test for the direct detection of Norovirus GI/GII RNA from stool specimens obtained from symptomatic patients.

The purpose of this study is to establish the diagnostic accuracy of ARIES Norovirus Assay.

DETAILED DESCRIPTION:
The ARIES Norovirus Assay is a real-time polymerase chain reaction (PCR) based qualitative in vitro diagnostic test for the direct detection of Norovirus GI/GII RNA from stool specimens obtained from symptomatic patients.

The objective is to establish the diagnostic accuracy of the ARIES Norovirus assay through a multi-site, method comparison on prospectively collected leftover, stool specimens. Diagnostic accuracy will be expressed in terms of clinical sensitivity (or positive agreement) and specificity (or negative agreement)

ELIGIBILITY:
Inclusion Criteria:

* The specimen is from a patient with symptoms of acute gastroenteritis.
* The specimen is from a male or female subject who was either hospitalized, admitted to a hospital emergency department or visiting an outpatient clinic.
* The subject's specimen is an unpreserved, unformed (liquid or soft) stool submitted for testing at the site.

Exclusion Criteria:

* The specimen is from an individual with known and documented non-infectious conditions such as ulcerative colitis, irritable bowel syndrome and/or Crohn's disease
* The specimen was not properly collected, transported, processed or stored according to the instructions provided by the sponsor.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All comers
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy will be expressed in terms of clinical sensitivity (or positive agreement) and specificity (or negative agreement). | Within the first year of sample collection
  Accuracy determinations (diagnostic sensitivity and specificity, positive and negative agreement) were based on the fraction of comparator positive (or negative) results which were also positive (or negative) by ARIES Norovirus Assay.

CONTACTS AND LOCATIONS:
Overall Officials: David Himsworth, Study Director — Luminex Corporation
Locations (5):
- United States (5):
  - UCLA, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Indiana Health, Indianapolis, Indiana
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Geisinger Medical Laboratories, Danville, Pennsylvania